CLINICAL TRIAL: NCT00706719
Title: A Randomized, Open-Label, Fixed Dose, Active-Control, Multi-Center Phase IIB Study to Evaluate Fertility in Men With Secondary Hypogonadism, Comparing Androxal® to a Topical Testosterone in Men Previously Treated With Topical Testosterone.
Brief Title: To Evaluate Sperm Parameters in Men With Secondary Hypogonadism Previously Treated With Topical Testosterone
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Repros Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZA-201
Record Dates: First submitted 2008-06-25; First posted 2008-06-27 (Estimated); Results first posted 2010-10-08 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-07

CONDITIONS: Secondary Hypogonadism
Keywords: Adult Onset Idiopathic Hypothalamic Hypogonadism (AIHH); Secondary hypogonadism; Semen volume; Sperm count; Sperm motility
MeSH Terms: conditions — Hypogonadism | interventions — Enclomiphene; Testosterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 25 mg Androxal no wash out (Experimental): 1 capsule daily for 6 months of 25 mg of Androxal in men without a 3 month wash out period
  Interventions: Drug: 25 mg Androxal
- Testim 1% (topical testosterone) (Active Comparator): Testim 1% Gel applied topically for 6 months
  Interventions: Drug: Testim 1%
- 25 mg Androxal wash out (Experimental): 1 x 25 mg Androxal capsule daily for 6 months in men with a previous 3 month washout period of topical testosterone
  Interventions: Drug: 25 mg Androxal

INTERVENTIONS:
Drug: 25 mg Androxal — 25 mg Androxal capsules, 1 capsule daily for 6 months
  Other Names: Enclomiphene citrate
  Arms: 25 mg Androxal no wash out; 25 mg Androxal wash out
Drug: Testim 1% — Testim 1% gel, dosage to be titrated according to manufacturer's instructions, once daily for 6 months
  Other Names: Topical testosterone
  Arms: Testim 1% (topical testosterone)

SUMMARY:
The study was designed to determine if Androxal® would affect sperm parameters (count, concentration, volume) in men with secondary hypogonadism who have been previously treated with topical testosterone.

DETAILED DESCRIPTION:
The study was designed to determine if Androxal® would affect sperm parameters (count, concentration, volume) in men with secondary hypogonadism who have been previously treated with topical testosterone. A maximum of twelve subjects per group were randomized to daily treatments of Androxal® or topical testosterone (Testim®) for six months. The protocol was later amended to include a treatment group who received Androxal after a 3 month wash out period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males between 21 and 60 years of age who have been diagnosed with AIHH.
* Subjects must have been treated with a topical testosterone replacement therapy (typically AndroGel® or Testim®) for at least 6 months at enrollment and for not more than 2 years.

Exclusion Criteria:

* A history of idiopathic infertility due to primary hypogonadism, testicular failure, Kallmann's syndrome or any other infertility condition.
* Subjects demonstrating any clinically significant medical condition rendering the subjects infertile or marginally fertile other than AIHH.
* Men with a history of, known, or suspected prostate disease not ruled out by a prostate biopsy, or a prostate specific antigen (PSA)>3.6 or clinical suspicion of current prostate disease.
* Men with a hematocrit in excess of 50 % or hemoglobin >17 g/dl

Ages: 21 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2008-06; Primary Completion 2009-07 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Wiehle, PhD, Study Director — Repros Therapeutics Inc.
Locations (2):
- United States (2):
  - University Urology Associates, New York, New York
  - MAZE Labs, Purchase, New York

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A Testim (Topical Testosterone): 1% Testim gel applied once daily
- Group B Androxal no Washout: 25 mg Androxal capsules once daily in men who have not previously washed out topical testosterone
- Group C Androxal With Wash Out: 25 mg capsules once daily in men who have previously had a 3 month wash out of topical testosterone
Period: Overall Study
Arm/Group | Group A Testim (Topical Testosterone) | Group B Androxal no Washout | Group C Androxal With Wash Out
Started | 5 | 7 | 5
Completed | 5 | 6 | 1
Not Completed | 0 | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Group A Testim: 1% Testim gel applied daily
- Group B Androxal no Wash Out: 25 mg Androxal 1 capsule per day in men who have not previously washed out topical testosterone for 3 months
- Group C Androxal Wash Out: 25 mg 1 capsule per day in men who have undergone a 3 month wash out period of topical testosterone
- Total: Total of all reporting groups
Arm/Group | Group A Testim | Group B Androxal no Wash Out | Group C Androxal Wash Out | Total
Number analyzed (Participants) | 5 | 7 | 5 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 7 | 5 | 17
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.4 (4.88) | 48.9 (8.99) | 56.4 (23.8) | 52.7 (7.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 5 | 7 | 5 | 17
Region of Enrollment [Number; unit: participants]
  United States | 5 | 7 | 5 | 17

OUTCOME MEASURES:

1. Primary Outcome: Sperm Concentration
Description: Total sperm concentration was measured.
Time Frame: Baseline, Month 3, Month 6, Follow-Up (Month 7)
Population: Subjects in Group A and B who completed the study. No analysis was performed for subjects in Group C because only 1 subject completed the study.
Measure: Mean (Standard Deviation); unit: millions sperm/mL
Arm/Group | Group A Testim | Group B Androxal no Wash Out
Number analyzed (Participants) | 5 | 6
millions sperm/mL
  Baseline | 0.54 (0.74) | 72.8 (92.7)
  Month 3 | 3.00 (5.20) | 182.6 (115.5)
  Month 6 | 23.14 (30.67) | 168.5 (92.9)
  Follow-Up (Month 7) | 21.03 (28.90) | 164.0 (71.2)
Statistical Analysis 1: Comparison: Group A Testim vs Group B Androxal no Wash Out; Comparison of Group A and B observed values at Baseline; Test type: Superiority or Other; p = 0.118, t-test, 2 sided
Statistical Analysis 2: Comparison: Group A Testim vs Group B Androxal no Wash Out; Comparison of Group A and B observed values at Month 3; Test type: Superiority or Other; p = 0.006, t-test, 2 sided
Statistical Analysis 3: Comparison: Group A Testim vs Group B Androxal no Wash Out; Comparison of Group A and B observed values at Month 6; Test type: Superiority or Other; p = 0.009, t-test, 2 sided
Statistical Analysis 4: Comparison: Group A Testim vs Group B Androxal no Wash Out; Comparison of Group A and B observed values at Follow-up (Month 7); Test type: Superiority or Other; p = 0.0024, t-test, 2 sided

2. Primary Outcome: Motile Total Sperm Count
Description: Motile total sperm count was measured.
Time Frame: Baseline, Month 3, Month 6, Follow-Up (Month 7)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millions sperm
Arm/Group | Group A Testim | Group B Androxal no Wash Out
Number analyzed (Participants) | 5 | 6
millions sperm
  Baseline | 0.3 (0.48) | 99.0 (159.6)
  Month 3 | 2.42 (5.41) | 214.7 (166.0)
  Month 6 | 40.4 (55.3) | 146.9 (120.0)
  Follow-Up (Month 7) | 38 (52.5) | 100.3 (103.8)
Statistical Analysis 1: Comparison: Group A Testim vs Group B Androxal no Wash Out; Comparison of Group A and B observed values at Baseline; Test type: Superiority or Other; p = 0.15, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Group A Testim vs Group B Androxal no Wash Out; Comparison of Group A and B observed values at Month 3; Test type: Superiority or Other; p = 0.0067, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Group A Testim vs Group B Androxal no Wash Out; Comparison of Group A and B observed values at Month 6; Test type: Superiority or Other; p = 0.10, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Group A Testim vs Group B Androxal no Wash Out; Comparison of Group A and B observed values at Follow-up (Month 7); Test type: Superiority or Other; p = 0.26, t-test, 2 sided

3. Primary Outcome: Semen Volume
Description: Semen volume was measured.
Time Frame: Baseline, Month 3, Month 6, Follow-Up (Month 7)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Group A Testim | Group B Androxal no Wash Out
Number analyzed (Participants) | 5 | 6
mL
  Baseline | 2.34 (1.43) | 2.23 (0.81)
  Month 3 | 2.88 (1.40) | 2.45 (1.31)
  Month 6 | 1.90 (1.03) | 2.48 (1.53)
  Follow-Up (Month 7) | 3.34 (0.83) | 2.40 (0.58)
Statistical Analysis 1: Comparison: Group A Testim vs Group B Androxal no Wash Out; Comparison of Group A and B observed values at Baseline; Test type: Superiority or Other; p = 0.880, t-test, 2 sided
Statistical Analysis 2: Comparison: Group A Testim vs Group B Androxal no Wash Out; Comparison of Group A and B observed values at Month 3; Test type: Superiority or Other; p = 0.612, t-test, 2 sided
Statistical Analysis 3: Comparison: Group A Testim vs Group B Androxal no Wash Out; Comparison of Group A and B observed values at Month 6; Test type: Superiority or Other; p = 0.488, t-test, 2 sided
Statistical Analysis 4: Comparison: Group A Testim vs Group B Androxal no Wash Out; Comparison of Group A and B observed values at Follow-up (Month 7); Test type: Superiority or Other; p = 0.054, t-test, 2 sided

4. Secondary Outcome: Luteinizing Hormone (LH) Levels
Description: LH levels were measured.
Time Frame: Baseline, Month 3, Month 6, Follow-Up (Month 7)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mIU/mL
Arm/Group | Group A Testim | Group B Androxal no Wash Out
Number analyzed (Participants) | 5 | 6
mIU/mL
  Baseline | 3.40 (2.14) | 2.92 (1.69)
  Month 3 | 0.88 (1.39) | 5.70 (3.22)
  Month 6 | 0.60 (0.58) | 6.12 (3.15)
  Follow-Up (Month 7) | 2.68 (0.48) | 2.47 (1.58)
Statistical Analysis 1: Comparison: Group A Testim vs Group B Androxal no Wash Out; Comparison of Group A and B observed values at Baseline; Test type: Superiority or Other; p = 0.705, t-test, 2 sided
Statistical Analysis 2: Comparison: Group A Testim vs Group B Androxal no Wash Out; Comparison of Group A and B observed values at Month 3; Test type: Superiority or Other; p = 0.013, t-test, 2 sided
Statistical Analysis 3: Comparison: Group A Testim vs Group B Androxal no Wash Out; Comparison of Group A and B observed values at Month 6; Test type: Superiority or Other; p = 0.004, t-test, 2 sided
Statistical Analysis 4: Comparison: Group A Testim vs Group B Androxal no Wash Out; Comparison of Group A and B observed values at Follow-up (Month 7); Test type: Superiority or Other; p = 0.808, t-test, 2 sided

5. Secondary Outcome: Follicle Stimulating Hormone (FSH) Levels
Description: FSH levels were measured.
Time Frame: Baseline, Month 3, Month 6, Follow-Up (Month 7)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mIU/mL
Arm/Group | Group A Testim | Group B Androxal no Wash Out
Number analyzed (Participants) | 5 | 6
mIU/mL
  Baseline | 3.38 (0.74) | 1.58 (0.74)
  Month 3 | 1.06 (1.12) | 4.53 (2.36)
  Month 6 | 0.9 (0.51) | 5.48 (2.46)
  Follow-Up (Month 7) | 3.6 (1.20) | 2.38 (0.95)
Statistical Analysis 1: Comparison: Group A Testim vs Group B Androxal no Wash Out; Comparison of Group A and B observed values at Baseline; Test type: Superiority or Other; p = 0.008, t-test, 2 sided
Statistical Analysis 2: Comparison: Group A Testim vs Group B Androxal no Wash Out; Comparison of Group A and B observed values at Month 3; Test type: Superiority or Other; p = 0.015, t-test, 2 sided
Statistical Analysis 3: Comparison: Group A Testim vs Group B Androxal no Wash Out; Comparison of Group A and B observed values at Month 6; Test type: Superiority or Other; p = 0.003, t-test, 2 sided
Statistical Analysis 4: Comparison: Group A Testim vs Group B Androxal no Wash Out; Comparison of Group A and B observed values at Follow-up (Month 7); Test type: Superiority or Other; p = 0.109, t-test, 2 sided

ADVERSE EVENTS:
Groups:
- Androxal Wash Out: 25 mg 1 capsule per day in men who have undergone a 3 month wash out period of topical testosterone
Arm/Group | Group A Testim | Group B Androxal no Wash Out | Androxal Wash Out
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/7 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 2/7 | 4/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A Testim (N=5) | Group B Androxal no Wash Out (N=7) | Androxal Wash Out (N=5)
diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
erythema (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1)
worsening depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
blurred vision (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
vasomotor flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other